CLINICAL TRIAL: NCT03348826
Title: Sodium Bicarbonate Injections for Restoration of Flow in a Central Venous Catheter (CVC/Hickman Catheter) or Peripherally Inserted Central Venous Catheter (PICC)
Brief Title: Study of Sodium Bicarbonate in Restoring Blocked Catheters
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No participants were enrolled
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SBI-FLOW
Record Dates: First submitted 2017-11-16; First posted 2017-11-21 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Cancer; Central Venous Catheterization
MeSH Terms: conditions — Neoplasms | interventions — Sodium Bicarbonate; Solutions; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alteplase then Sodium Bicarbonate (Experimental): Alteplase will first be administered to restore flow. If flow is not restored, then sodium bicarbonate will be administered.
  Interventions: Drug: Sodium Bicarbonate 8.4% Solution for Injection; Drug: Alteplase Injectable Solution
- Sodium Bicarbonate then Alteplase (Experimental): Sodium bicarbonate will first be administered to restore flow. If flow is not restored, then alteplase will be administered.
  Interventions: Drug: Sodium Bicarbonate 8.4% Solution for Injection; Drug: Alteplase Injectable Solution

INTERVENTIONS:
Drug: Sodium Bicarbonate 8.4% Solution for Injection — 3 mL injection into line with up to 2 injections administered
Drug: Alteplase Injectable Solution — 2 mL injection into line with up to 2 injections administered

SUMMARY:
This is a study looking at the use of sodium bicarbonate to restore the flow of blocked central line devices in patients with blood cancers.

Central line devices uses thin tubes that are placed into a vein in the body to give medicines, fluids, nutrients, blood products, etc.

Sometimes, the lines become blocked. The standard procedure to get the line working again is to use alteplase, a protein that dissolves blood clots. While blood clotting is one cause of a blocked line, other reasons included the formation of calcium deposits. Sodium bicarbonate is routinely used in the treatment of patients receiving chemotherapy. Sodium bicarbonate is a liquid drug which is capable of dissolving protein and calcium deposits.

This study will compare whether sodium bicarbonate works just as well as alteplase to recover the function of a blocked line.

ELIGIBILITY:
Inclusion Criteria:

* Hematology patients with indwelling CVC/PICC line.
* Patients continuing to receive chemotherapy treatment for consolidation, intensification and maintenance regimens in hematological malignancies such as in acute leukemia, lymphoma, myelodysplastic syndrome, supportive care measures using blood products, ongoing anti-infective treatments, and nutrition.
* Patients whose CVC/PICC line becomes obstructed during routine care are being identified and presented to attending physician and pharmacist.
* Mechanical obstruction having been ruled out by visual inspection and manipulation of the patient's posture or extremities or both.

Exclusion Criteria:

* Patients with hemodialysis line occlusions
* Anyone with documentation of prior history of alteplase allergy or hypersensitivity reactions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2021-09-02 (Estimated)

PRIMARY OUTCOMES:
Successful clearance rate of sodium bicarbonate | 3 hours
Successful clearance rate of alteplase | 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Mark Minden, M.D., Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No